CLINICAL TRIAL: NCT05663164
Title: Effect of Thiamine on Serum Glucagon And Reactive Oxygen Species (ROS) in Perioperative Stress Response
Brief Title: Effect of Thiamine on Serum Glucagon And Reactive Oxygen Species (ROS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, Bastian Lubis, Head of Intensive Care Unit, Universitas Sumatera Utara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2022-11-23; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Sepsis; Thiamine Deficiency
Keywords: thiamine; sepsis; glucagon; ROS; Perioperative Stress Response
MeSH Terms: conditions — Sepsis; Thiamine Deficiency | interventions — Folic Acid; Thiamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Vitamin B1 (Experimental): Vitamin B1 (thiamine) 100mg every 6 hours x 3-days
  Interventions: Drug: Vitamin B
- Drug: Normal saline (Placebo Comparator): Normal saline (0.9% NaCl solution) volume to match all components
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin B — vitamin B1 (100mg) will be diluted in 50 ml 0.9% NACL(normal saline) and administered IV every 6 hours for 3 days
  Other Names: Thiamine
  Arms: Experimental: Vitamin B1
Drug: Placebo — Normal saline (0.9% NaCl solution) volume to match all components
  Other Names: Normal saline
  Arms: Drug: Normal saline

SUMMARY:
This research is a clinical trial with a Randomized Controlled Trial (RCT) design. The purpose is to identify the effect of intravenous thiamine administration compared to normal saline placebo on glucagon levels and ROS levels in patients undergoing general anesthesia surgery

DETAILED DESCRIPTION:
Surgery may increase postoperative cortisol and blood glucose levels. Changes in normal metabolic patterns due to surgery stimulate gluconeogenesis, glycogenolysis, proteolysis, lipolysis, and cytogenesis. These result in hyperglycemia and ketosis conditions. Surgery and anesthesia lead to an immunosuppressive effect. Increased secretion of proinflammatory cytokines may also occur after the surgery.

Besides an increase in cortisol levels, surgery can also increase cytokine response and ROS production in patients who have undergone surgery under general anesthesia after 72 hours. ROS production can also be a useful indicator in assessing the severity of surgical trauma.

In surgical procedures, there is an acute increase in reactive oxidative stress (ROS). This occurs when ischemia is followed by reperfusion. ROS can trigger tissue injury seen in transplantation (liver and heart), the release of aortic clamps during abdominal and thoracic aortic surgery, the release of limb tourniquets during orthopedic surgery, and reperfusion during and after cardiopulmonary bypass. There is a thiamine deficiency in 20% of patients treated in the intensive care unit (ICU). Thiamine deficiency is a source of lactic acidosis that does not seem in severe sepsis and septic shock. An imbalance between the formation and removal of free radicals causes a pathological condition called oxidative stress. However, the human body uses antioxidants to suppress these free radicals. One of the antioxidants that can reduce oxidative stress is thiamine. Previous studies proved this finding. Thiamine has also been able to significantly prevent the expression of inflammatory cytokines and chemokines, depending on NF-B induced by thromboxane and PGI2 synthase.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years who undergo surgery under general anesthesia
* ASA physical statuses 1 and 2
* Sepsis

Exclusion Criteria:

* Refuse to participate
* Diabetes mellitus, experience shock sepsis or lactic acidosis
* Have a history of hypersensitivity (allergy) to thiamine
* Thiamine deficiency
* Take immunomodulatory drugs, antiplatelet or anticoagulants surgery duration > 6 hours, and thiamin regularly
* They experience massive bleeding and receive blood transfusions preoperatively, intraoperatively, or postoperatively

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Glucagon Level | On day 3 (at approximately 72 hours) after the first study drug dose
  a hormone that your pancreas makes to help regulate your blood glucose (sugar) levels
ROS Level | On day 3 (at approximately 72 hours) after the first study drug dose
  Reactive species is the common term for both free radicals and reactive oxygen species (ROS), which include radicals, such as superoxide radical anion and hydroxyl radical, and nonradicals, such as hydrogen peroxide

CONTACTS AND LOCATIONS:
Overall Officials: Bastian Lubis, Dr, Principal Investigator — Faculty of Medicine Universitas Sumatera Utara
Locations (1):
- Faculty of Medicine Universitas Sumatera Utara, Medan, North Sumatra, Indonesia

REFERENCES:
- [Background] Cusack B, Buggy DJ. Anaesthesia, analgesia, and the surgical stress response. BJA Educ. 2020 Sep;20(9):321-328. doi: 10.1016/j.bjae.2020.04.006. Epub 2020 Jul 21. No abstract available. PMID 33456967
- [Background] Prete A, Yan Q, Al-Tarrah K, Akturk HK, Prokop LJ, Alahdab F, Foster MA, Lord JM, Karavitaki N, Wass JA, Murad MH, Arlt W, Bancos I. The cortisol stress response induced by surgery: A systematic review and meta-analysis. Clin Endocrinol (Oxf). 2018 Nov;89(5):554-567. doi: 10.1111/cen.13820. Epub 2018 Aug 23. PMID 30047158
- [Background] Davis G, Fayfman M, Reyes-Umpierrez D, Hafeez S, Pasquel FJ, Vellanki P, Haw JS, Peng L, Jacobs S, Umpierrez GE. Stress hyperglycemia in general surgery: Why should we care? J Diabetes Complications. 2018 Mar;32(3):305-309. doi: 10.1016/j.jdiacomp.2017.11.010. Epub 2017 Nov 29. PMID 29273446
- [Background] Sudhakaran S, Surani SR. Guidelines for Perioperative Management of the Diabetic Patient. Surg Res Pract. 2015;2015:284063. doi: 10.1155/2015/284063. Epub 2015 May 19. PMID 26078998
- [Background] Hazell AS, Faim S, Wertheimer G, Silva VR, Marques CS. The impact of oxidative stress in thiamine deficiency: a multifactorial targeting issue. Neurochem Int. 2013 Apr;62(5):796-802. doi: 10.1016/j.neuint.2013.01.009. Epub 2013 Jan 18. PMID 23333339
- [Background] Costa NA, Gut AL, de Souza Dorna M, Pimentel JA, Cozzolino SM, Azevedo PS, Fernandes AA, Zornoff LA, de Paiva SA, Minicucci MF. Corrigendum to "serum thiamine concentration and oxidative stress as predictors of mortality in patients with septic shock" [J Crit care 2014;29(2):249-52]. J Crit Care. 2016 Dec;36:311. doi: 10.1016/j.jcrc.2016.07.001. Epub 2016 Jul 10. No abstract available. PMID 27810062
- [Background] Luong KV, Nguyen LT. The impact of thiamine treatment in the diabetes mellitus. J Clin Med Res. 2012 Jun;4(3):153-60. doi: 10.4021/jocmr890w. Epub 2012 May 15. PMID 22719800
- [Background] Karkabounas S, Papadopoulos N, Anastasiadou C, Gubili C, Peschos D, Daskalou T, Fikioris N, Simos YV, Kontargiris E, Gianakopoulos X, Ragos V, Chatzidimitriou M. Effects of alpha-Lipoic Acid, Carnosine, and Thiamine Supplementation in Obese Patients with Type 2 Diabetes Mellitus: A Randomized, Double-Blind Study. J Med Food. 2018 Dec;21(12):1197-1203. doi: 10.1089/jmf.2018.0007. Epub 2018 Oct 11. PMID 30311825
- [Background] Lubis B, Lelo A, Amelia P, Prima A. The Effect of Thiamine, Ascorbic Acid, and the Combination of Them on the Levels of Matrix Metalloproteinase-9 (MMP-9) and Tissue Inhibitor of Matrix Metalloproteinase-1 (TIMP-1) in Sepsis Patients. Infect Drug Resist. 2022 Sep 30;15:5741-5751. doi: 10.2147/IDR.S378523. eCollection 2022. PMID 36204393